CLINICAL TRIAL: NCT01292707
Title: A Cluster-randomised Trial of Health Worker and Community Interventions to Improve Adherence to National Guidelines for the Use of ACTs in Tanzania
Brief Title: A Cluster-randomised Trial of Interventions to Improve Antimalarial Prescribing With Malaria Tests
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Ministry of Health, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ACTc TACT
Record Dates: First submitted 2011-01-28; First posted 2011-02-09 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Malaria
Keywords: malaria; rdt; fever; treatment
MeSH Terms: conditions — Malaria; Rhabdoid Tumor; Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Prescribing staff in control facilities will receive the standard package of RDT training that is being provided by NMCP in Tanzania
  Interventions: Behavioral: Control
- HW (Active Comparator): Prescribing staff in the intervention facilities will receive the same package of nationally-approved training in RDT use as will be provided to prescribers in control facilities. Following this, prescribers in the intervention facilities will be invited to participate in 3 small group training modules delivered in an interactive style lasting approximately 11/2 hours, with one session repeated between the 6th and 7th month of the trial.
  Interventions: Behavioral: HW
- HWC (Active Comparator): The health worker-community arm will receive the same intervention as the health workers arm but with the addition of an intervention aimed at patients. This will consist of community sensitisation, clinic posters and providing a leaflet to each RDT-tested patient or caretaker giving details of the test and the corresponding treatment provided.
  Interventions: Behavioral: HWC

INTERVENTIONS:
Behavioral: Control — Standard national training
  Arms: Control
Behavioral: HW — Prescribing staff in the intervention facilities will receive the same package of nationally-approved training in RDT use as will be provided to prescribers in control facilities. Following this, prescribers in the intervention facilities will be invited to participate in 3 small group training modules delivered in an interactive style lasting approximately 11/2 hours, with one session repeated between the 6th and 7th month of the trial
  Arms: HW
Behavioral: HWC — The health worker-community arm will receive the same intervention as the health workers arm but with the addition of an intervention aimed at patients. This will consist of community sensitisation, clinic posters and providing a leaflet to each RDT-tested patient or caretaker giving details of the test and the corresponding treatment provided.
  Arms: HWC

SUMMARY:
Background.

Overdiagnosis of malaria is widespread in health facilities throughout Africa, a situation that is unsustainable given the relatively high cost of artemisinin combination therapy (ACTs) compared to older antimalarials. In addition it often denies patients treatment for their actual illness and generates unreliable data for health planners. For these reasons the National Malaria Control Programme introduced revised guidelines for malaria diagnosis and treatment in 2006 restricting the recommendation for antimalarial treatment in patients over the age of 5 years to those with a positive blood slide or malaria rapid diagnostic tests (RDTs) result. To support this, RDTs will be introduced into primary care health facilities in Tanzania starting in 2009.

The high accuracy of current rapid diagnostic tests (RDTs) provides the potential for a cost-effective solution to the problem of malaria overdiagnosis. However, RDTs with revised guidelines to restrict malaria diagnoses to RDT-positive patients have been unsuccessful unless accompanied by unsustainable levels of supervision and training.

Primary objective.

To conduct a trial of interventions directed at prescribers or prescribers and communities compared to control groups to improve adherence to national guidelines for prescription of antimalarial treatment when supported by RDTs in primary health care facilities in NE Tanzania.

Methods

All 60 participating health facilities will receive RDTs and basic training in their use and a copy of current NMCP/MOH guidelines for each prescribing staff member. A health worker intervention arm will, in addition, receive workplace-based interactive training and messages from senior staff A health worker-community arm will receive the same training as the health worker arm and in addition leaflets will be provided to RDT-tested patients providing information on the test and the treatment given. All training materials will be approved by NMCP in Tanzania as being consistent with current national guidelines but with the addition that prescribers will be asked to follow RDT results in prescribing for patients of any age This policy is in line with the most recent revision to WHO guidelines and is supported by NMCP in Tanzania.

Study outcomes will be recorded through a 40% (2 days per week) exit survey of patients. Anthropological and economics studies will assess the costs and acceptability of interventions.

ELIGIBILITY:
Health Facility Inclusion criteria:

* Located in lowland Muheza, adjoining wards of Handeni, or any area of Moshi Rural Districts
* Health facilities that are registered with the District Health Authority
* Receives Government supplies of ALu and qualifies for RDT supply
* Agrees to exclusive use of RDT for routine diagnosis of first consultations for possible malaria
* Accessible by 4-wd vehicle throughout the year.
* Availability of data on proportion of consultations diagnosed with malaria in 2008 (or earliest available year)

Health Facility Exclusion:

* Presence of other research in the immediate area where study procedures could bias outcomes in either study.
* Fewer than 500 cases per year were reported in 2005 or 2006.

Patient Inclusion:

* All patients with non-severe illness in first consultations.
* Patient Exclusion
* Patients who have been referred to the next level of care
* Patient refuses consent to exit survey
* Follow-up consultations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a non-severe non-malarial illness prescribed a recommended antimalarial drug in a new consultation. | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Reyburn, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Joint Malaria Programme, Moshi, Kilimanjaro, Tanzania

REFERENCES:
- [Derived] Leurent B, Reyburn H, Muro F, Mbakilwa H, Schellenberg D. Monitoring patient care through health facility exit interviews: an assessment of the Hawthorne effect in a trial of adherence to malaria treatment guidelines in Tanzania. BMC Infect Dis. 2016 Feb 3;16:59. doi: 10.1186/s12879-016-1362-0. PMID 26842751
- [Derived] Cundill B, Mbakilwa H, Chandler CI, Mtove G, Mtei F, Willetts A, Foster E, Muro F, Mwinyishehe R, Mandike R, Olomi R, Whitty CJ, Reyburn H. Prescriber and patient-oriented behavioural interventions to improve use of malaria rapid diagnostic tests in Tanzania: facility-based cluster randomised trial. BMC Med. 2015 May 15;13:118. doi: 10.1186/s12916-015-0346-z. PMID 25980737
- [Derived] Chandler CI, Meta J, Ponzo C, Nasuwa F, Kessy J, Mbakilwa H, Haaland A, Reyburn H. The development of effective behaviour change interventions to support the use of malaria rapid diagnostic tests by Tanzanian clinicians. Implement Sci. 2014 Jun 26;9:83. doi: 10.1186/1748-5908-9-83. PMID 24969367